CLINICAL TRIAL: NCT05674019
Title: Analyse Des Sillons Corticaux Par IRM morphométrique : développement de Biomarqueurs neurodéveloppementaux Des Troubles Bipolaires
Brief Title: MOrphometric MRI Analysis of Cortical Sulci: Development of NEurodevelopmental Biomarkers of Bipolar Disorder.
Acronym: NEMO-Bipolar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RCAPHM21_0440
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Neurodevelopemental Group Non-neurodevelopmental Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurodevelopmental Group (Experimental): The volunteer presents at least 2 of 12 neurodevelopmental crieria
  Interventions: Other: MRI exam
- Non-neurodevelopmental Group (Active Comparator): The volunteer does not present any of the 12 neurodevelopmental crieria
  Interventions: Other: MRI exam

INTERVENTIONS:
Other: MRI exam — Brain MRI Morphometric exam

SUMMARY:
Given the phenotypic heterogeneity of bipolar disorder, it seems essential to propose new methodologies to improve the stratification of this pathology in order to describe more homogeneous groups of patients. In this perspective, the neurodevelopmental hypothesis of bipolar disorder seems promising. Brain sulcation is an indirect marker of neurodevelopmental processes. The objective of the study is to highlight sulcal variations between a group of bipolar patients with a neurodevelopmental phenotype (ND) and a group of bipolar subjects without a ND phenotype. A sulcation marker (GPR56) will also be measured from patient blood samples. In order to carry out this project we would like to include 120 participants for a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

For the "neurodevelopmental" group :

The volunteer has at least 2 of the 12 neurodevelopmental criteria

For the "non-neurodevelopmental" group The volunteer does not present any of the 12 neurodevelopmental criteria

List of the 12 neurodevelopmental criteria :

1. The volunteer had at birth a paternal age ≥ 40 years
2. The volunteer had at birth a maternal age ≥ 35 years
3. The volunteer was born by cesarean section
4. The volunteer had a history of perinatal infection
5. The volunteer has a history of generalized anxiety disorder that began before the age of 16 (≤ 15 years)
6. The volunteer has a history of an eating disorder that began before the age of 16 (≤ 15 years)
7. The volunteer has a history of a substance use disorder (excluding tobacco) as described in the DSM-5 prior to age 16 (≤ 15 years)
8. The volunteer has a learning disability or "dys" disorder as defined in the DSM-5 or number of repeats > 2
9. The volunteer has a history of trauma assessed as severe by the CTQ self-assessment questionnaire
10. The volunteer has symptoms suggestive of Attention Deficit Hyperactivity Disorder (WURS score > 46)
11. The volunteer has a history of psychotic features during episodes.
12. The volunteer has an early age of onset of bipolar disorder at an age below 18 years.

Exclusion Criteria:

* Serious symptomatic or unstable physiological or medical condition (including pregnancy)
* History of stable or non-stable psychiatric illness, schizophrenia or any other condition that may interfere with bipolar disorder
* History of comorbid autism spectrum disorder
* History of severe head injury (GCS<8 at time of injury)
* Neurological disorder affecting central nervous system function
* Moderate to severe substance use disorder (>=4/11 as defined in the DSM-5) with the exception of tobacco use disorder
* Under court protection or guardianship
* Unable to give the volunteer informed information, or the volunteer refuses to sign the consent form
* Insufficient command of the French language to complete the assessments
* Has a contraindication to MRI

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2025-01-14 (Estimated); Study Completion 2025-01-14 (Estimated)

PRIMARY OUTCOMES:
Diifference in the occurrence of sulcal pits allowing to discriminate between a group of bipolar patients presenting a neurodevelopmental phenotype and a group of bipolar patients not presenting this phenotype. | 24 months
  Patients are identified in the neurodevelopmental group following a list of 12 criteria (0 criterion = non neurodevelopmental, at leat 2 criteria = neurodevelopmental)

SECONDARY OUTCOMES:
The depth and number of sulcal pits to differentiate a group of bipolar patients with a neurodevelopmental phenotype from a group of bipolar patients without this phenotype. | 24 months
  Patients are identified in the neurodevelopmental group following a list of 12 criteria (0 criterion = non neurodevelopmental, at leat 2 criteria = neurodevelopmental)
The demonstration of correlations between different scores used in the clinic that may be related to neurodevelopmental manifestations of bipolar disorder (scales: WURS, minor neurological signs scale) and the number of sulcal-pits. | 24 months
  Patients are identified in the neurodevelopmental group following a list of 12 criteria (0 criterion = non neurodevelopmental, at leat 2 criteria = neurodevelopmental)
The blood level of GRP56 messenger RNA measured in whole blood by quantitative PCR to differentiate a group of bipolar patients with a neurodevelopmental phenotype and a group of bipolar patients without this phenotype | 24 months
  Patients are identified in the neurodevelopmental group following a list of 12 criteria (0 criterion = non neurodevelopmental, at leat 2 criteria = neurodevelopmental)
Genetic polymorphisms of GPR56 to differentiate between a group of bipolar patients with a neurodevelopmental phenotype and a group of bipolar patients without this phenotype | 24 months
  Patients are identified in the neurodevelopmental group following a list of 12 criteria (0 criterion = non neurodevelopmental, at leat 2 criteria = neurodevelopmental)
Protein quantification of the circulating fraction of GP56 in plasma and serum to differentiate a group of bipolar patients with a neurodevelopmental phenotype from a group of bipolar patients without this phenotype. | 24 months
  Patients are identified in the neurodevelopmental group following a list of 12 criteria (0 criterion = non neurodevelopmental, at leat 2 criteria = neurodevelopmental)

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — AP-HM

IPD SHARING:
Plan to Share IPD: No